CLINICAL TRIAL: NCT02468167
Title: Comparison of Endoscopic Cyanoacrylate Injection Versus Balloon-occluded Retrograde Transvenous Obliteration in the Management of Acute Gastric Variceal Bleeding
Brief Title: Acute Gastric Variceal Bleeding: Endoscopic Treatment Versus BRTO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, luo xuefeng, MD, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BRTO-NBCA-AB
Record Dates: First submitted 2015-06-03; First posted 2015-06-10 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Gastric Varices
MeSH Terms: conditions — Esophageal and Gastric Varices | interventions — Enbucrilate; Polidocanol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BRTO (Active Comparator): Balloon-occluded retrograde transvenous obliteration
  Interventions: Procedure: Balloon-occluded retrograde transvenous obliteration; Drug: Lauromacrogol
- NBCA (Active Comparator): Endoscopic cyanoacrylate injection
  Interventions: Procedure: Endoscopic cyanoacrylate injection; Drug: N-butyl-2-cyanoacrylate

INTERVENTIONS:
Procedure: Balloon-occluded retrograde transvenous obliteration — Balloon-occluded retrograde transvenous obliteration
  Arms: BRTO
Procedure: Endoscopic cyanoacrylate injection — Endoscopic cyanoacrylate injection
  Arms: NBCA
Drug: N-butyl-2-cyanoacrylate
  Arms: NBCA
Drug: Lauromacrogol
  Arms: BRTO

SUMMARY:
The purpose of this study is to study the efficacy of endoscopic cyanoacrylate injection versus balloon-occluded retrograde transvenous obliteration in the management of acute gastric bleeding.

ELIGIBILITY:
Inclusion Criteria:

1. Cirrhosis
2. Active bleeding from gastric varices (GOV2 or IGV1)
3. Presence of gastrorenal shunt

Exclusion Criteria:

1. Previous pharmacologic therapy combined with endoscopic treatment to prevent rebleeding
2. Previous use of TIPS or surgical shunt
3. Non-cirrhotic portal hypertension
4. Contraindications to cyanoacrylate injection or BRTO
5. Portal cavernoma
6. Hepatorenal syndrome
7. Proven malignancy including hepatocellular carcinoma
8. End-stage renal disease under renal replacement therapy;
9. Cardiorespiratory failure
10. Pregnancy or patients not giving informed consent for endoscopic procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
The number of participants with failure to control acute bleeding or failure to prevent clinically significant variceal rebleeding within 1 year after enrollment | 1 year

SECONDARY OUTCOMES:
Mortality rate | 3 years
Eradication rate of gastric varices | 3 years
Number of participants with increase or decrease in the size of gastric varices | 3 years
Number of participants with appearance or worsening of new oesophageal varices | 3 years
Number of participants with appearance or worsening of portal hypertensive gastropathy | 3 years
Number of participants with appearance or worsening of ascites | 3 years
Number of participants with complication | 3 years
Average in-hospital stay | 3 years
Cost of treatment | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuan, China